CLINICAL TRIAL: NCT04416971
Title: Clinical Values of Mature Fistulas in Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Bo Shen, Principal Investigator, Shanghai Zhongshan Hospital
Other Study IDs: Mature Fistulas
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Hemodialysis Access Failure; Hemodialysis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mature AVF: Patients initiate HD with mature AVF.
  Interventions: Procedure: AVF puncture
- immature AVF: Patients initiate HD with immature AVF.
  Interventions: Procedure: AVF puncture

INTERVENTIONS:
Procedure: AVF puncture — For patients with mature/immature AVF on HD initiation, AVF puncture will be conducted.

SUMMARY:
The arteriovenous fistula (AVF) is the preferred vascular access for hemodialysis(HD), and fistula-first is the general recommendation for all HD patients. But in clinical practice in China, quite a few patients start HD before AVF maturation due to various situations. Whether HD initiation with mature AVF will influence the patency and complications is controversial. This study is aim to compare the AVF patency in incident HD patients with mature or immature AVF on HD initiation, and to compare other clinical outcomes, including abandonment without use, infection, and other AVF complications occurrence.

ELIGIBILITY:
Inclusion Criteria:

* underwent initial upper-extremity AVF creation for incident HD at Zhongshan Hospital, Fudan University

Exclusion Criteria:

* with malignancies
* not followed-up at Zhongshan Hospital, Fudan University

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * aged 18 years and older
  * underwent initial upper-extremity AVF creation for incident HD at our hospital
  * divided into mature/immature AVF groups according to the AVF status on HD initiation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
AVF patency | June 2020 to June 2021
  A functional AVF was defined as allowing at least six adequate HD sessions without any AVF-related complications. Primary AVF patency was defined as the interval from HD initiation via a functional AVF to any intervention designed for maintenance or reestablishment of AVF function, AVF failure, or study end, whichever occurred first, and secondary AVF patency was defined as the interval from HD initiation via an AVF until the termination of HD via AVF due to any cause, regardless of the number of subsequent interventions.

SECONDARY OUTCOMES:
Abandonment without use, infection, and other complications of AVF creation. | June 2020 to June 2021
  Abandonment without use, infection, and other complications of AVF creation.

CONTACTS AND LOCATIONS:
Overall Officials: bo shen, MD, Principal Investigator — Fudan University
Locations (1):
- No.180, Fenglin Road, Xuhui District, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No